CLINICAL TRIAL: NCT04739059
Title: An Open-label Study to Evaluate the Long-term Safety and Efficacy of CSL312 (Garadacimab) in the Prophylactic Treatment of Hereditary Angioedema
Brief Title: Long-term Safety and Efficacy of CSL312 (Garadacimab) in the Prophylactic Treatment of Hereditary Angioedema Attacks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSL312_3002; 2020-003918-12 (EudraCT Number)
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CSL312 (Experimental): Fully human immunoglobulin G subclass 4/lambda recombinant inhibitor monoclonal antibody administered subcutaneously
  Interventions: Biological: CSL312

INTERVENTIONS:
Biological: CSL312 — Fully human immunoglobulin G subclass 4/lambda recombinant inhibitor monoclonal antibody
  Other Names: Factor XIIa inhibitor monoclonal antibody; garadacimab

SUMMARY:
This phase 3b study will evaluate long-term safety and efficacy of CSL312 (also known as garadacimab) when administered subcutaneously (SC)

ELIGIBILITY:
Inclusion Criteria:

* - Males and females aged ≥ 12 years
* - Diagnosed with clinically confirmed C1-INH HAE
* - Experienced ≥ 3 HAE attacks during the 3 months before Screening
* - Participated in the Run-in Period for at least 1 month (CSL312-naïve subjects only)
* - Experienced at least an average of 1 HAE attack per month during the Run-in Period

Exclusion Criteria:

* - Concomitant diagnosis of another form of angioedema, such as idiopathic or acquired angioedema or recurrent angioedema associated with urticaria
* - Use of C1-INH products, androgens, antifibrinolytics or other small molecule medications for routine prophylaxis against HAE attacks at least 2 weeks before the first day of the Run-in Period
* - Use of monoclonal antibodies such as lanadelumab (Takhzyro®) 3 months before the first day of the Run-in Period.
* - Female subjects use estrogen-containing oral contraceptives or hormone replacement therapy within 4 weeks prior to screening
* - Female or male subjects who are fertile and sexually active not using or not willing to use an acceptable method of contraception to avoid pregnancy during the study and for 30 days after receipt of the last dose of CSL312
* - Pregnant, breastfeeding, or not willing to cease breastfeeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment emergent adverse events (TEAEs) | Up to 45 months
Percentage of subjects with TEAEs | Up to 45 months
TEAEs rates per injection | Up to 45 months
TEAEs rates per subject year | Up to 45 months

SECONDARY OUTCOMES:
The time-normalized number (per month and year) of Hereditary Angioedema (HAE attacks) for the entire study | Up to 43 months
The percentage reduction and the number of subjects experiencing at least ≥ 50% ≥ 70%, ≥ 90 or equal to 100% (attack free) reduction in the time-normalized number of HAE attacks on Treatment compared to Run-in Period | Up to 43 months
The time-normalized number (per month and year) of HAE attacks requiring on-demand treatment in subjects on treatment | Up to 43 months
The time-normalized number (per month and year) of moderate and/or severe HAE attacks in subjects on treatment | Up to 43 months
Number and percentage of subjects rating their response to therapy as good or excellent | Up to 43 months
The number and percentage of subjects experiencing TEAEs | Up to 45 months
The number and percentage of subjects experiencing adverse events of special interest (AESIs) | Up to 45 months
The number and percentage of subjects experiencing serious adverse events (SAEs), including deaths | Up to 45 months
The number and percentage of subjects experiencing CSL312 induced anti-CSL312 antibodies | Up to 45 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (44):
- United States (11):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Research Solutions of Arizona, Litchfield Park, Arizona
  - Medical Research of Arizona, Scottsdale, Arizona
  - Little Rock Allergy & Asthma Clinic, Little Rock, Arkansas
  - Donald S. Levy M.D., Orange, California
  - Raffi Tachdjian MD, Inc., Santa Monica, California
  - Allergy & Asthma Clinical Research, Walnut Creek, California
  - Institute for Asthma and Allergy PC, Chevy Chase, Maryland
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - PennState Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - AARA Research Center, Dallas, Texas
- Australia (3):
  - Campbelltown Hospital / Western Sydney University, Campbelltown, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Department of Clinical Immunology, Murdoch, Western Australia
- Canada (5):
  - University of Alberta - Research Transition Facility, Edmonton, Alberta
  - McMaster University, Hamilton, Ontario
  - Ottawa Allergy Research Corp, Ottawa, Ontario
  - Gordon Sussman Clinical Research, Toronto, Ontario
  - Montreal Clinical Research Institute, Montreal, Quebec
- Czechia (2):
  - University hospital St. Anna Ustav klinicke imunologie a alergologie, Fakultní nemocnice u sv. Anny v Brně, Brno
  - University Hospital Motol, Prague
- Germany (4):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt
  - Johannes Gutenberg-Universität KöR, Hautklinik und Poliklinik der Universitätsmedizin, Clinical Research Center, Mainz
  - HZRM Haemophilie Zentrum Rhein Main GmbH, Mörfelden-Walldorf
- The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong
- Semmelweis Egyetem Altalanos Orvostudományi Kar Belgyógyászati és Hematológiai Klinika, Budapest, Hungary
- Barzilai University Medical Center, Ashkelon, Israel
- Japan (10):
  - Koga Community Hospital, Shizuoka, Daikakuji Yaizu-shi
  - Mie University Hospital, Mie, Edobashi, Tsu-shi
  - Juntendo University Hospital, Tokyo, Hongo Bunkyo-ku
  - Saitama Medical Center, Saitama, Kamoda Kawagoe-shi
  - St. Marianna University School of Medicine Hospital, Kanagawa, Kawasaki-shi
  - Clover Hospital, Kanagawa, Kugenumaishigami, Fujisawa-shi
  - Saiyu Soka Hospital, Saitama, Matsubara Soka-shi
  - National Hospital Organization Disaster Medical Center, Tokyo, Midoricho, Tachikawa-shi
  - Saga University Hospital, Saga, Nebeshima, Saga-shi
  - Local Incorporated Administrative Agency Osaka City Hospital Organization Osaka City General Hospital, Miyakojima-ku, Osaka-shi
- Amsterdam UMC, location AMC, Amsterdam, Netherlands
- Auckland City Hospital, Grafton, Auckland, New Zealand
- NRC Institute of Immunology FMBA Russia, Moscow, Russia
- Spain (2):
  - Hospital Universitari General de La Vall d'Hebron, Barcelona
  - Hospital Gregorio Marañón, Servicio de Alergia, Madrid
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.